CLINICAL TRIAL: NCT05446714
Title: Evaluation of Three Types of Rapid Maxillary Expanders (Conventional, Hybrid, And MSE) on Maxilla in Adolescent A Randomized Clinical Trial - CBCT Study
Brief Title: Evaluation of the Effect of Three Types of Rapid Maxillary Expanders (Conventional, Hybrid and MSE)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Mohamed Abdelrhman Shendy Abdelrhman, Clinical professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 775/220; Ahmed (Other: AlAzhar); lecturer (Registry Identifier: Ahmed Abo Elnour)
Record Dates: First submitted 2022-06-20; First posted 2022-07-07 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Maxillary Retrusion; Nasal Airway Obstruction
MeSH Terms: conditions — Retrognathia; Nasal Obstruction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional hyrax (Active Comparator): CH 4 BANDS for expansion of maxilla and observation improvement of the air way
  Interventions: Device: CH 4 band
- Hybrid hyrax (Active Comparator): HH 2 BANDS for expansion of maxilla and observation improvement of the air way
  Interventions: Device: HH 2 bands
- Maxillary skeletal expander (Active Comparator): MSE 2 BANDS AND 4 for expansion of maxilla and observation improvement of the air way
  Interventions: Device: MSE 2 bands and 4

INTERVENTIONS:
Device: CH 4 band — expansion of maxilla and observation improvement of the air way
  Other Names: rapid palatal expansion; Orthodontic rapid maxillary expansion
  Arms: conventional hyrax
Device: HH 2 bands — expansion of maxilla and observation improvement of the air way
  Arms: Hybrid hyrax
Device: MSE 2 bands and 4 — expansion of maxilla and observation improvement of the air way
  Arms: Maxillary skeletal expander

SUMMARY:
Aim of the study: To compare radiographically the morphometric changes in the nasal airway after using three types of rapid maxillary expansion (RME) conventional hyrax (CH), hybrid hyrax (HH) and maxillary skeletal expander (MSE) using cone beam computed tomography (CBCT).

DETAILED DESCRIPTION:
Abstract Aim of the study: To compare radiographically the morphometric changes in the nasal airway after using three types of rapid maxillary expansion (RME) conventional hyrax (CH), hybrid hyrax (HH) and maxillary skeletal expander (MSE) using cone beam computed tomography (CBCT).

Material and Methods: A total sample of thirty CBCT of patients presented with constricted maxilla with mean age of 14±3Y was randomized in to three groups. Group 1 CH, group 2 HH and group 3 MSE.

CBCT records were taken before(T1) and after six months (T2) of RME; the Airway was segmented and quantified using software (version 5.3.4.39USA).

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering maxillary collapse with a skeletal background
* Patients with unilateral or bilateral posterior crossbite.
* Patients with reduced or average anterior face height.
* Patients with no periodontal disease.
* Patients with good oral hygiene and general health.
* No systemic diseases that may affect bone quality or interfere with orthodontic treatment.
* Patients with erupted maxillary permanent first molars and premolars.
* Patients with no previous orthodontic treatment.

Exclusion Criteria:

* previous treatment
* syndromes
* cleft lip and palate

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 54 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2023-11-19 (Actual); Study Completion 2025-06-20 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shendy, Principal Investigator — Al-Azhar University
Locations (1):
- Cairo, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
CBCT Measurements
Supporting Information: Study Protocol, ICF
Time Frame: 6 months
Access Criteria: Constricted maxilla

REFERENCES:
- [Background] Gracco A, Malaguti A, Lombardo L, Mazzoli A, Raffaeli R. Palatal volume following rapid maxillary expansion in mixed dentition. Angle Orthod. 2010 Jan;80(1):153-9. doi: 10.2319/010407-7.1. PMID 19852655
- [Result] Lagravere MO, Major PW, Flores-Mir C. Long-term skeletal changes with rapid maxillary expansion: a systematic review. Angle Orthod. 2005 Nov;75(6):1046-52. doi: 10.1043/0003-3219(2005)75[1046:LSCWRM]2.0.CO;2. PMID 16448254

RESULTS

PARTICIPANT FLOW:
Recruitment Details: orthodontic department al-azhar university
Pre-assignment Details: * Patients suffering maxillary collapse with a skeletal background
  * Patients with unilateral or bilateral posterior crossbite.
  * Patients with reduced or average anterior face height.
  * Patients with no periodontal disease.
  * Patients with good oral hygiene and general health.6- No systemic diseases that may affect bone quality or interfere with orthodontic treatment.
  * Patients with erupted maxillary permanent first molars and premolars.
Period: Overall Study
Arm/Group | Conventional Hyrax | Hybrid Hyrax | Maxillary Skeletal Expander
Started | 18 | 18 | 18
Completed | 15 (interruption=3) | 15 (broken appliance) | 16 (failure of miniscrews)
Not Completed | 3 | 3 | 2
Not completed — Lost to Follow-up | 1 | 3 | 2
Not completed — Protocol Violation | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Hyrax | Hybrid Hyrax | Maxillary Skeletal Expander | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Categorical [Count of Participants; unit: Participants] — Population: dropout due to bad oral hygiene
  Participants
    s: <=18 years | 6 | 6 | 6 | 18
    s: Between 18 and 65 years | 6 | 7 | 6 | 19
    s: >=65 years | 6 | 5 | 6 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.50 (1.04) | 13.96 (1.21) | 13.81 (0.98) | 14.09 (1.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 17
  Male | 13 | 12 | 12 | 37
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Molar Distance:
Description: distance in milimeter from mesiolingual cusp of upper first molar in one side to mesiolingual cusp of upper first molar in the other CBCT Measurements software
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Conventional Hyrax | Hybrid Hyrax | Maxillary Skeletal Expander
Number analyzed (Participants) | 15 | 15 | 16
mm | 43.55 (1.97) | 44.79 (4.27) | 42.14 (3.25)

2. Secondary Outcome: Molar Inclination
Description: amount of degree of Molar inclination change before and after maxillary expansion which measured from the long axis of upper first molar to palatal plane by CBCT Evaluation
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Conventional Hyrax | Hybrid Hyrax | Maxillary Skeletal Expander
Number analyzed (Participants) | 15 | 15 | 16
mm | 5.66 (1.52) | 4.85 (2.10) | 2.08 (1.30)

3. Secondary Outcome: Maxillary Width
Description: amount of maxillary width changes by CBCT Evaluation
Time Frame: 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Temporomandibular Joint
Description: CBCT Evaluation
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Conventional Hyrax | Hybrid Hyrax | Maxillary Skeletal Expander
All-Cause Mortality (participants affected / at risk) | 15/18 | 15/18 | 16/18
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 1/18
Other Adverse Events (participants affected / at risk) | 1/18 | 1/18 | 2/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Hyrax (N=18) | Hybrid Hyrax (N=18) | Maxillary Skeletal Expander (N=18)
metabolism (Metabolism and nutrition disorders) | 1 (2) | 1 (1) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conventional Hyrax (N=18) | Hybrid Hyrax (N=18) | Maxillary Skeletal Expander (N=18)
cardiac (Cardiac disorders) | 1 (1) | 1 (2) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-28): https://cdn.clinicaltrials.gov/large-docs/14/NCT05446714/Prot_002.pdf
  • Statistical Analysis Plan (2024-05-14): https://cdn.clinicaltrials.gov/large-docs/14/NCT05446714/SAP_003.pdf